CLINICAL TRIAL: NCT07383857
Title: PULSAR Radiotherapy Plus Anti-PD-1 Therapy in Metastatic Abdominopelvic Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhen Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhen Zhang, Director, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2502314-15
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Radiation: pulsed radiotherapy

INTERVENTIONS:
Radiation: pulsed radiotherapy — All enrolled participants will receive pulsed radiotherapy (PULSAR)

SUMMARY:
This study evaluates hypofractionated radiotherapy combined with PD-1 inhibitor-based systemic therapy in patients with metastatic solid tumors. Eligible patients will be enrolled into three cohorts according to tumor type: metastatic hepatocellular carcinoma, metastatic renal cell carcinoma, and metastatic urothelial carcinoma. The study aims to assess the safety and therapeutic efficacy of combining localized radiotherapy with immunotherapy, with or without cohort-specific systemic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of enrollment, with no restriction on sex.
2. Histologically, cytologically, or radiologically confirmed metastatic abdominopelvic malignancy, including hepatocellular carcinoma, renal cell carcinoma, or urothelial carcinoma.
3. No more than 10 metastatic lesions, and the radiotherapy treatment plan indicates that radiotherapy can be safely delivered.
4. At least one measurable lesion is present.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Determined by a multidisciplinary team (MDT) to require active antitumor treatment.
7. Adequate bone marrow, liver, renal, and coagulation function as demonstrated by laboratory tests performed within 7 days prior to the first dose of study treatment; no blood transfusion, blood products, granulocyte colony-stimulating factor (G-CSF), or other hematopoietic growth factors are permitted within 7 days prior to laboratory testing.
8. Voluntary participation with written informed consent provided, and willingness to comply with the study treatment protocol and scheduled visits.

Exclusion Criteria:

1. Absolute neutrophil count (ANC) <1.5 × 10⁹/L, or platelet count <100 × 10⁹/L (or <80 × 10⁹/L in patients with liver metastases), or hemoglobin <9 g/dL; blood transfusion within 2 weeks prior to enrollment to meet eligibility criteria is not permitted.
2. Serum total bilirubin >1.5 × the upper limit of normal (ULN), or >2.5 × ULN in patients with liver metastases.
3. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 × ULN, or >5 × ULN in patients with liver metastases.
4. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m².
5. Clinically significant electrolyte abnormalities as determined by the investigator.
6. Active gastrointestinal diseases, including but not limited to gastric or duodenal ulcers, ulcerative colitis, or active bleeding from unresected tumors; or other conditions judged by the investigator to carry a risk of gastrointestinal bleeding or perforation; or a history of gastrointestinal perforation or fistula that has not fully healed after surgical treatment.
7. History of arterial thrombosis or deep vein thrombosis within 6 months prior to enrollment, or evidence or history of bleeding tendency within 2 months prior to enrollment, regardless of severity.
8. Stroke or transient ischemic attack within 12 months prior to enrollment.
9. Significant cardiac disease within 6 months prior to enrollment, including congestive heart failure, acute myocardial infarction, severe or unstable angina, or coronary artery bypass grafting; or New York Heart Association (NYHA) class II or higher heart failure; or left ventricular ejection fraction (LVEF) <50%.
10. Presence of a clinically detectable second primary malignancy at screening, or a history of another malignancy within the past 5 years, except for adequately treated early-stage non-melanoma skin cancer, carcinoma in situ of the cervix, superficial bladder cancer (non-muscle-invasive tumors, carcinoma in situ, or T1 tumors), or early-stage thyroid cancer.
11. Known clinically significant liver disease, including but not limited to hepatitis B virus (HBV) infection with positive HBV DNA (≥1 × 10⁴ IU/mL), hepatitis C virus (HCV) infection with positive HCV RNA (≥1 × 10³ IU/mL), or cirrhosis.
12. Pregnant or breastfeeding women, women of childbearing potential with a positive pregnancy test prior to first dosing, or participants (or their partners) unwilling to use effective contraception during the study period.
13. Any clinical or laboratory abnormality or compliance issue that, in the investigator's judgment, makes the participant unsuitable for participation in this study.
14. Presence of severe psychological or psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China